CLINICAL TRIAL: NCT05053516
Title: Development and Effectiveness Evaluation of the Standardized Training Program for Social Workers for Drug Treatment Based on Industry Needs
Brief Title: the Standardized Training Program for Social Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: JDu-009
Record Dates: First submitted 2021-06-19; First posted 2021-09-22 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-06

CONDITIONS: Social Workers; Educational Problems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the intervention group (Other): The intervention group will participate in the training program of this study, while the control group will receive the existing routine training program.
  Interventions: Other: A standardized training program for social workers
- the control group (Other): The intervention group will participate in the training program of this study, while the control group will receive the existing routine training program.
  Interventions: Other: A standardized training program for social workers

INTERVENTIONS:
Other: A standardized training program for social workers — A standardized training program for social workers who work with drug addicts / drug users based on industry needs

SUMMARY:
Now, there are few researches on the ability of social workers who work with drug addicts / drug users in China, and the sample size is small and the content is not deep enough.The existing studies suggest that the professional knowledge and ability of social workers who work with drug addicts / drug users are insufficient and the vocational training is not standardized. On the other hand, the ability of social workers who work with drug addicts / drug users workers is related to the effectiveness of anti-drug in communities. So the large sample survey will help to understand the current working status and working ability of social workers who work with drug addicts / drug users in China.The development of the standardized training programs for social workers who work with drug addicts / drug users can improve the professional knowledge and ability of anti-drug social workers, so as to better help community drug rehabilitation personnel and finally reduce the relapse rate.

ELIGIBILITY:
Inclusion Criteria:

- aged between 20 and 65;no gender limitation;those who agree to participate in the study and sign the informed consent.

Exclusion Criteria:

- inability to use online training.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive competency assessment | 3 months
  Comprehensive competency assessment Focus interview: It is planned to recruit 8 anti-drug social workers for focus interviews.Adopt the minimum sample principle, and stop recruiting when new objects cannot provide new information.Outline of interviews: Is the time, content of the training reasonable? Whether the training has achieved the desired effect? If not, what are the shortcomings?

IPD SHARING:
Plan to Share IPD: No